CLINICAL TRIAL: NCT06558552
Title: Comparison of the Efficacy of Posterior Tibial Nerve Neuromodulation and Extracorporeal Shock Wave Therapy for Heel Spur: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halil Ibrahim Altun (Other)
Responsible Party: Sponsor-Investigator, Halil Ibrahim Altun, pain specialist, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: heelspur
Record Dates: First submitted 2024-08-12; First posted 2024-08-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neuromodulation of the Posterior Tibial Nerve in the Heel Spur (Epin Calcanei) (Other)
  Interventions: Other: transcutaneous pulsed radiofrequency
- extracorporeal shock wave therapy (ESWT) (Other)
  Interventions: Other: extracorporeal shock wave therapy (ESWT)'

INTERVENTIONS:
Other: transcutaneous pulsed radiofrequency — Instead of invasive application of PRF directly to the lesion area or nerve, transcutaneous pulsed radiofrequency (TCPRF) is applied noninvasively.
  Arms: Neuromodulation of the Posterior Tibial Nerve in the Heel Spur (Epin Calcanei)
Other: extracorporeal shock wave therapy (ESWT)' — A shock wave is created together with sound and pressure waves. Changes at the cellular level with the shock wave include increased collagen production, increased blood flow in the applied area, acceleration of wound healing and cellular proliferation.
  Arms: extracorporeal shock wave therapy (ESWT)

SUMMARY:
Heel pain is an important clinical condition that impairs patients' quality of life and causes loss of workforce. Heel spurs are one of the most important causes of heel pain. Heel spur, often plantar fascia calcaneus It is seen at the site of attachment to the tuberosity and is plantar It develops secondary to microtrauma to the calcaneus following inflammation of the fascia , and over time, an organized bone protrusion called a spur forms in the same area . Plantar in patients with heel spurs It is often accompanied by fasciitis . Heel spurs are more common in women. It increases with increasing age due to mechanical trauma to the heel. Its incidence is not clearly known . In its etiology, age, gender, obesity, foot structure that disrupts biomechanics, rheumatological and metabolic diseases, and trauma come to the fore .

Nonsteroids in the treatment of heel spurs There are treatment options such as anti-inflammatory drugs (NSAIDs), other analgesics, exercise, splints and orthoses, shoe insoles and pads, corticosteroid injections into the spur area and extracorporeal shock wave therapy (ESWT). There are a limited number of studies in which pulse radiofrequency (PRF) and injection were applied to the posterior tibial nerve, which senses the region , and conventional or pulse radiofrequency was successfully applied to the lesion area .

ESWT is a non-invasive method. A shock wave is created together with sound and pressure waves. Changes at the cellular level with the shock wave include increased collagen production, increased blood flow in the applied area, acceleration of wound healing and cellular proliferation. In ESWT, radial and focal waves are applied depending on the tissue depth. patellar tendinopathy , plantar fasciitis , myositis It is an effective and reliable method that is frequently used in the treatment of ossificans , lateral epicondylitis , iliotibial band syndrome, many tendinopathies and heel spurs .

PRF is a newer neuromodulation method than conventional radiofrequency. It increases c-fos gene expression at the cellular level in neurons without causing destructive damage to the nerve , and A-delta and C fibers are affected. algogenic neuromediators decrease, endogenous opioids such as Dynorphin , Enkephalin and Endorphin increase, thus reducing pain.

DETAILED DESCRIPTION:
The study will include 48 patients between the ages of 18 and 65, diagnosed with heel spurs, who meet the inclusion and exclusion criteria in the Algology and PMR (Physical medicine and rehabilitation) departments of Kanuni Sultan Süleyman Training and Research Hospital, between sep 2024 and apr 2025 (Standard effect As a result of the power analysis, it was deemed appropriate to include at least 22 cases in each group with a power of 80% and a margin of error of 0.84 . According to this result, a total of 48 patients will be included in the study, taking into account the losses ). Randomization will be done using a randomization program to divide patients into two groups and assign a number to each patient.

The power analysis, it was deemed appropriate to include at least 22 cases in each group , with a standard effect size of 0.84, with 80% power and 5% margin of error . According to this result, a total of 48 patients will be included in the study, taking into account losses .) The posterior tibial nerve will be performed by the same algologist . Patients will be monitored standardly (Noninvasive blood pressure, pulse oximeter, electrocardiogram) and will be performed in the supine position at TCPRF . For TCPRF, a 45*98 mm diameter transcutaneous electrode (FIAB SPA, Italy ) will be used. Electrode medial at ankle level It will be placed posterior to the malleolus , in the posterior tibial nerve trace accompanying the artery after palpation of the posterior tibial artery . TCPRF will be applied for 8 minutes at 80 volts, 2 Hz, 20 ms . The process will be repeated 3 times with a one-week interval.

To the control group with the radial ESWT device. Vibrolith An Orto® brand electro- pneumatic , extracorporeal shock wave therapy device will be used. It will be applied by the same physiotherapist with at least 10 years of experience in the field. Sick It will be in the prone position and ESWT will be applied to the spur area as a radial type shock wave . The process will be repeated 3 times with a one-week interval. Sessions will be applied with 10 Hz frequency, 2000 beats, 2.5 bar intensity.

Patient evaluation and results will be made by another algologist (FAE) who is unaware of the type of treatment. Demographic data of the patients, body mass index (BMI), symptom duration, additional diseases, medical treatments, the side where the procedure was performed, rest and activity Numeric Rating Scale -11 ( NRS) and Foot function index ( Foot ) function index , FFI) will be recorded before the procedure and in the 1st and 3rd months after the procedure. NRS-11 is an 11-point numerical scale in which patients can evaluate their pain between 0 (no pain) and 10 (the most severe pain they have ever felt in their life) . FFI is a validated scale consisting of 23 questions in total, including 3 subgroups : pain, disability and activity limitation .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65,
* Patients diagnosed with calcaneus spur and epin calcaneus in radiological imaging with anamnesis, clinical and physical examination
* Patients who signed the voluntary consent form

Exclusion Criteria:

* Patients who have undergone interventional procedures for heel spurs in the last 6 months,
* Morbidly obese patients (BMI>35 kg/m2),
* Patients with advanced decompensated heart failure and pacemakers,
* Patients with known transcutaneous pad allergy, patients with skin infection in the area where ESWT was performed or pads were attached,
* Patients with metal implants,
* Patients with circulatory disorders and lesions,
* Patients who cannot communicate and cannot be positioned,
* Patients with bleeding disorders, patients with severe psychosis and progressive neurological deficits and muscle diseases,
* and pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
foot function index | four months

CONTACTS AND LOCATIONS:
Overall Officials: halil ibrahim altun, specialist, Principal Investigator — Kanuni Sultan Süleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No